CLINICAL TRIAL: NCT07235059
Title: A Participant- and Investigator--Blinded, Placebo- Controlled, Randomized, Multipart, Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of OJR520 in Healthy Volunteers and Participants With Chronic Kidney Disease
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of OJR520 in Healthy Volunteers and Participants With Chronic Kidney Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: COJR520A12101; 2025-520978-18 (Other: EU Trial (CTIS) number)
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease
Keywords: OJR520; safety and tolerability; PK; PD; healthy volunteers; first in human; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Part A: OJR520 dose A1 (Experimental): Participants will receive OJR520 dose level A1.
  Interventions: Drug: OJR520
- Part A: OJR520 dose A2 (Experimental): Participants will receive OJR520 dose level A2.
  Interventions: Drug: OJR520
- Part A: OJR520 dose A3 (Experimental): Participants will receive OJR520 dose level A3.
  Interventions: Drug: OJR520
- Part A: OJR520 dose A4 (Experimental): Participants will receive OJR520 dose level A4.
  Interventions: Drug: OJR520
- Part A: OJR520 dose A5 (Experimental): Participants will receive OJR520 dose level A5.
  Interventions: Drug: OJR520
- Part A: OJR520 dose A6 (Experimental): Participants will receive OJR520 dose level A6.
  Interventions: Drug: OJR520
- Part B: OJR520 dose B1 (Experimental): Participants will receive OJR520 dose level B1.
  Interventions: Drug: OJR520
- Part B: OJR520 dose B2 (Experimental): Participants will receive OJR520 dose level B2.
  Interventions: Drug: OJR520
- Part B: OJR520 dose B3 (Experimental): Participants will receive OJR520 dose level B3.
  Interventions: Drug: OJR520
- Part B: OJR520 dose B4 (Experimental): Participants will receive OJR520 dose level B4.
  Interventions: Drug: OJR520
- Part C: OJR520 dose C1 (Experimental): Participants will receive OJR520 dose level C1.
  Interventions: Drug: OJR520
- Part C: OJR520 dose C2 (Experimental): Participants will receive OJR520 dose level C2.
  Interventions: Drug: OJR520
- Part C: OJR520 dose C3 (Experimental): Participants will receive OJR520 dose level C3.
  Interventions: Drug: OJR520
- Part C: OJR520 dose C4 (Experimental): Participants will receive OJR520 dose level C4.
  Interventions: Drug: OJR520
- Part A: Placebo (Placebo Comparator): Participants will receive the matching placebo.
  Interventions: Other: Placebo
- Part B: Placebo (Placebo Comparator): Participants will receive the matching placebo.
  Interventions: Other: Placebo
- Part C: Placebo (Placebo Comparator): Participants will receive the matching placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: OJR520 — Participants will receive OJR520 in different dose levels.
  Arms: Part A: OJR520 dose A1; Part A: OJR520 dose A2; Part A: OJR520 dose A3; Part A: OJR520 dose A4; Part A: OJR520 dose A5; Part A: OJR520 dose A6; Part B: OJR520 dose B1; Part B: OJR520 dose B2; Part B: OJR520 dose B3; Part B: OJR520 dose B4; Part C: OJR520 dose C1; Part C: OJR520 dose C2; Part C: OJR520 dose C3; Part C: OJR520 dose C4
Other: Placebo — Participants will receive OJR520 matching placebo.
  Arms: Part A: Placebo; Part B: Placebo; Part C: Placebo

SUMMARY:
The purpose of this first-in-human (FIH) study is to evaluate safety, tolerability, pharmacokinetic (PK) of OJR520.

DETAILED DESCRIPTION:
This is a three-part randomized, participant- and investigator blinded, placebo-controlled, multi-center, sequential study: single ascending dose (SAD) in healthy volunteers (HV), SAD in participants with chronic kidney disease (CKD) or diabetic chronic kidney disease (DKD) and multiple ascending dose (MAD) in participants with CKD or DKD.

ELIGIBILITY:
Inclusion Criteria:

Able to provide written informed consent before any assessment is performed.

Part A (HV):

• Healthy male and female participants in good health as determined by past medical history, physical examination, vital signs, 12-lead ECG, and laboratory tests at screening and baseline within the normal range.

Parts B & C (CKD)

• Male and female participants 18 to 65 years of age.

Exclusion Criteria:

* Women of childbearing potential.
* Sexually active males unwilling to use contraception.

Part A (HV):

* Clinically significant abnormal blood pressure, defined as SBP <90 mmHg or >140 mmHg or DBP <55 mmHg or >95 mmHg.
* Abnormal resting HR, defined as <45 bpm or >90 bpm.

Part B & C (CKD)

* History of, or currently active, significant illness or medical disorders including, but not limited to, cancer (except for non-melanoma skin cancer), heart failure NYHA III-IV, heart rhythm abnormalities (e.g., atrial fibrillation, sick sinus syndrome, permanent pacemaker), CKD due to autoimmune disease, kidney transplant, dialysis or any other disease the investigator believes may preclude the participant from participating in the this study.
* Clinically significant aortic stenosis or mitral insufficiency as identified via echocardiography.
* History of myocardial infarction (MI), stroke, coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI), or transient ischemic attack (TIA).

Other protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-07-19 (Estimated); Study Completion 2027-07-19 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse events (AEs) and Serious Adverse events (SAEs) | From Day 1 (Part A) until Day 71 (Part C)
  Incidence and severity of AEs and SAEs by treatment group, including changes in vital signs, electrocardiograms (ECGs) and laboratory results qualifying and reported as AEs.

SECONDARY OUTCOMES:
Maximum Observed Blood Concentrations (Cmax) | From pre-dose Day 1 (Part A) until Day 71 (Part C)
  Cmax is the maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration (mass x volume-1).
Time to reach maximum plasma concentration (Tmax) | From pre-dose Day 1 (Part A) until Day 71 (Part C)
  Tmax is the time to reach maximum (peak) drug concentration after single-dose administration (time).
Area under plasma concentration-time curve (AUClast) | From pre-dose Day 1 (Part A) until Day 71 (Part C)
  AUClast is the area under the plasma concentration-time curve from time zero to the time of last quantifiable concentration (tlast).
Area under the plasma concentration-time curve (AUC[0-inf]) | From pre-dose Day 1 (Part A) until Day 71 (Part C)
  The AUC[0-inf] from time zero extrapolated to infinity (mass x time x volume-1).
Terminal elimination half-life (T1/2) | From pre-dose Day 1 (Part A) until Day 71 (Part C)
  T1/2 is the elimination half-life associated with the terminal slope.
Apparent plasma clearance (CL/F) | From pre-dose Day 1 (Part A) until Day 71 (Part C)
  CL/F is the apparent total body clearance of drug from plasma following extravascular administration.
Apparent volume of distribution during terminal elimination phase (Vz/F) | From pre-dose Day 1 (Part A) until Day 71 (Part C)
  Vz/F is the apparent volume of distribution during terminal elimination phase following extravascular administration.
Drug accumulation ratio (Racc) | Part C: From pre-dose Day 1 until Day 71
  The ratio of accumulation of drug between the first and last dose, only for MAD part of the study.
Area under plasma concentration-time curve (AUCtau) | Part C: From pre-dose Day 1 until Day 71
  The AUC calculated to the end of a dosing interval (tau) (amount x time x volume-1) only for MAD part of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences Sea View, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No